CLINICAL TRIAL: NCT02462694
Title: High Risk Suicidal Behavior in Veterans - Assessment of Predictors and Efficacy of Dialectical Behavior Therapy
Brief Title: High Risk Suicidal Behavior in Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bronx Veterans Medical Research Foundation, Inc (Other)
Responsible Party: Principal Investigator, Marianne Goodman, Marianne Goodman, MD, Bronx Veterans Medical Research Foundation, Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOO-09-073
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide | interventions — Dialectical Behavior Therapy; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment as Usual (Active Comparator): Treatment as usual (TAU): Standard psychological, psychopharmacology and case management services
  Interventions: Behavioral: Treatment As Usual
- Dialectical Behavior Therapy (Experimental): Standard Dialectical Behavior Therapy (DBT): weekly individual sessions, skills training group and telephone coaching as needed
  Interventions: Behavioral: Dialectical Behavior Therapy

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy — Dialectical Behavior Therapy is an empirically validated treatment approach emphasizing the role of emotion regulation in the treatment of suicidal and self-destructive behaviors in BPD
  Arms: Dialectical Behavior Therapy
Behavioral: Treatment As Usual — TAU for these subjects involves close tracking by the Suicide Prevention Coordinator and treatment by their individual team of clinicians. Additionally, a support group with psychoeducation about suicide prevention will be offered as part of TAU
  Arms: Treatment as Usual

SUMMARY:
Suicide is a pressing problem in the US military, with evidence of increased risk for suicide particularly among soldiers serving in Iraq and Afghanistan. To date, there are very few studies that empirically evaluate treatment efficacy to prevent suicide. One treatment that has been shown empirically to decrease suicidal behavior is Dialectical Behavioral Therapy (DBT), although these studies have been limited to patients with borderline personality disorder (BPD). The current proposal aims to examine the efficacy of DBT in reducing suicidal behavior more broadly in a diagnostically heterogeneous group of veterans with high risk suicidal behavior. One of the difficulties in doing research in suicide prevention is that serious suicidal behavior is a relatively rare event, and alone is not a satisfactory target for treatment studies. It is extremely important, therefore, to identify intermediate symptoms that are closely associated with high risk suicidal behaviors, as targets for treatment. One critical area our proposal addresses is validating new treatment models for suicide in veterans; DBT has been empirically validated to reduce suicidal behavior in individuals with BPD, but has not been tested more broadly to target suicidal behaviors. The second critical area which our proposal addresses is exploring new suicide risk assessment measures. While the investigators do not specifically propose to develop new screening tools, the investigators do propose to identify potentially important domains that specifically differentiate ill high risk suicide veterans from low risk. This information will be useful in future efforts to modify the DBT approach to be more effective for the broader diagnostic group of high risk suicidal veterans.

DETAILED DESCRIPTION:
This project proposes two related studies. The first project is a randomized clinical trial of 120 veterans identified with high-risk suicidal behavior comparing the efficacy of DBT vs. treatment as usual (TAU) on suicidal behavior as a primary outcome measure. A second aim of the present project is to examine group differences between 200 300 veterans at high risk for suicide and 200 veterans at low risk in a variety of symptom domains. The goal of this will be to identify symptoms associated with suicidal behavior that can be used as secondary and exploratory outcome measures for DBT. The investigators will assess symptom domains including mood and substance use that have been associated with suicidal behavior by previous research and validate those in our veteran population by comparing symptoms in low vs. high risk veterans recently discharged from the James J Peters VAMC (JJPVA) psychiatric inpatient unit. In addition, the investigators will explore indices of interpersonal function and measure features that have some evidence of offering protection from suicide, which could be viewed as resilience factors. A particular emphasis of the present project is to characterize the nature of the interpersonal dysfunction in high risk individuals, as there exists very good evidence that social isolation, or a lack of a sense of "belonging" puts people at particularly high risk for suicide, in particular in a military sample. The investigators intend to assess the impact of DBT vs. TAU on these symptom domains in addition to their impact on suicidal behavior.

The subject population for both projects will be veterans identified on a "high risk" suicide list at the James J. Peters VAMC; veterans are so identified by the suicide coordinator because of a recent inpatient hospitalization involving high-risk suicidal behavior. Priority will be given to OEF/OIF veterans. In order to identify symptoms associated with high risk suicidal behavior, the investigators will examine symptoms domains in our high risk subjects and contrast them with a comparison group of veterans recently discharged from the psychiatric inpatient service or treated in the outpatient mental health department at the James J Peters VA Medical Center with no history of high-risk suicidal behaviors (low risk veterans). Groups will be matched with respect to age and gender. For this project, the investigators will include veterans with a variety of diagnoses, including post-traumatic stress disorder (PTSD), substance abuse, affective disorders, personality disorders, and anxiety disorders. The investigators will exclude subjects with current psychosis or cognitive impairment as these symptoms would prevent appropriate engagement in DBT. Patients from the high-risk suicide list will be eligible to participate in a six month DBT treatment study and will be randomized to full DBT vs. TAU. Both groups will have psychopharmacological management by their outpatient psychiatrist and be able to participate in standard ancillary outpatient clinical offerings (e.g. AA, sleep group). Both treatment groups will be assessed at baseline, at the 6 month treatment completion mark, as well as follow-up time points including one year and eighteen months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Veterans between the ages of 18 and 65
2. Able to give consent
3. Recent admission to psychiatric inpatient unit (6B)

Exclusion Criteria:

1. Lifetime or current diagnosis of schizophrenia or other psychotic disorder; current psychosis from affective disorder
2. IQ<80
3. Current evidence or history of significant organic brain impairment, including stroke, CNS tumor, demyelinating disease, severe head trauma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2010-04; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Counting of suicidal events | 6 months
  Utilizing the The Columbia Suicide Severity Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Goodman, MD, Principal Investigator — James J. Peters Veterans Affairs Medical Center

REFERENCES:
- [Derived] Goodman M, Banthin D, Blair NJ, Mascitelli KA, Wilsnack J, Chen J, Messenger JW, Perez-Rodriguez MM, Triebwasser J, Koenigsberg HW, Goetz RR, Hazlett EA, New AS. A Randomized Trial of Dialectical Behavior Therapy in High-Risk Suicidal Veterans. J Clin Psychiatry. 2016 Dec;77(12):e1591-e1600. doi: 10.4088/JCP.15m10235. PMID 27780335